CLINICAL TRIAL: NCT01404156
Title: PreOperative Treatment With chEmotheRapy or chemoRAdiatioN in esophaGeal or gastroEsophageal adenocaRcinoma
Brief Title: Preoperative Chemotherapy vs. Chemoradiation in Esophageal / GEJ Adenocarcinoma
Acronym: POWERRANGER
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. Gordon Buduhan (Other)
Collaborators: CancerCare Manitoba (Other); University of Toronto (Other); London Health Sciences Centre (Other)
Responsible Party: Sponsor-Investigator, Dr. Gordon Buduhan, MD MSc FRCSC Associate Professor of Surgery Section of Thoracic Surgery,, CancerCare Manitoba
Organization: CancerCare Manitoba (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDHA 174431-7
Record Dates: First submitted 2011-07-26; First posted 2011-07-27 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer; Adenocarcinoma, Esophageal; Adenocarcinoma, Gastroesophageal Junction
Keywords: Esophageal cancer; Neoadjuvant; Chemotherapy; Chemoradiation; Surgery; Esophagectomy; Adenocarcinoma; Gastroesophageal
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Adenocarcinoma | interventions — Capecitabine; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neoadjuvant Chemotherapy (Active Comparator): NEOADJUVANT CHEMOTHERAPY (OPTION of CHEMO REGIMEN 1 or 2)
  1) FLOT - Four x 14 day cycles FLOT preoperatively and 4 cycles postoperatively (within 4-10 weeks after surgery): 5-Fluorouracil 2600 mg/m², day 1 IV every 14 days Leucovorin 200 mg/m², day 1, IV., every 14 days Oxaliplatin 85 mg/m², day 1, IV, every 14 days Docetaxel 50mg/m2, day 1, IV, every 14 days
  2) ECF / ECX - Three x 21-day cycles ECF preoperatively and 3 cycles postoperatively (within 4-10 weeks after surgery): Epirubicin (50 mg/m²,mg per square meter of body-surface area) by intravenous bolus on day 1 IV Cisplatin: 60 mg/m², mg per square meter intravenously with hydration on day 1 IV 5-Fluorouracil: 200 mg/m², mg per square meter daily for 21 days by continuous intravenous infusionIV infusion 5-FU may be substituted with Capecitabine (Xeloda) 625mg/m2 PO BID (ECX)
  Interventions: Drug: (Epirubicin Cisplatin 5-Fluorouracil / Xeloda) OR 5-Fluorouracil Leucovorin Oxaliplatin Docetaxel
- Neoadjuvant Chemoradiation (Experimental): 1) -carboplatin and paclitaxel given on days 1, 8, 15, 22 and 29
  * paclitaxel: 50 mg / m2 IV over 1 hour
  * carboplatin: dosed to an area under the curve of 2, by Calvert formula, as a 1 hour IV infusion Radiation Therapy Concurrent radiation therapy will begin within 24 hours of initiation of chemotherapy for patients randomized to chemoradiation treatment.
    1. Dose specifications:
       1. Phase 1: Total radiation prescription dose 45 Gy given in 25 fractions of 1.8 Gy per fraction, 5 fractions / week, one treatment / day, starting on the first day of first cycle of chemotherapy.
       2. Phase 2: (GTV only) Boost is not mandatory and up to the discretion of radiation oncologist. Total radiation prescription dose 5.4 Gy given in 3 fractions of 1.8 Gy per fraction, 5 fractions / week, one treatment.
  Interventions: Other: Carboplatin paclitaxel plus concurrent radiotherapy

INTERVENTIONS:
Drug: (Epirubicin Cisplatin 5-Fluorouracil / Xeloda) OR 5-Fluorouracil Leucovorin Oxaliplatin Docetaxel — NEOADJUVANT CHEMOTHERAPY (OPTION of CHEMO REGIMEN 1 or 2)
  1) FLOT - Four x 14 day cycles FLOT preoperatively and 4 cycles postoperatively (within 4-10 weeks after surgery): 5-Fluorouracil 2600 mg/m², day 1 IV every 14 days Leucovorin 200 mg/m², day 1, IV., every 14 days Oxaliplatin 85 mg/m², day 1, IV, every 14 days Docetaxel 50mg/m2, day 1, IV, every 14 days
  2) ECF / ECX - Three x 21-day cycles ECF preoperatively and 3 cycles postoperatively (within 4-10 weeks after surgery): Epirubicin (50 mg/m²,mg per square meter of body-surface area) by intravenous bolus on day 1 IV Cisplatin: 60 mg/m², mg per square meter intravenously with hydration on day 1 IV 5-Fluorouracil: 200 mg/m², mg per square meter daily for 21 days by continuous IV infusion 5-FU may be substituted with Capecitabine (Xeloda) 625mg/m2, PO BID (ECX)
  Other Names: ECF/ECX or FLOT
  Arms: Neoadjuvant Chemotherapy
Other: Carboplatin paclitaxel plus concurrent radiotherapy — 5 cycles carboplatin and paclitaxel given on days 1, 8, 15, 22 and 29 preoperatively:
  * paclitaxel: 50 mg / m2 IV over 1 hour
  * carboplatin: dosed to an area under the curve of 2, by Calvert formula, as a 1 hour IV infusion
  Radiation Therapy Concurrent radiation therapy will begin within 24 hours of initiation of chemotherapy for patients randomized to chemoradiation treatment.
  1. Dose specifications:
  1. Phase 1: Total radiation prescription dose 45 Gy given in 25 fractions of 1.8 Gy per fraction, 5 fractions / week, one treatment / day, starting on the first day of first cycle of chemotherapy. This total radiation dose option is acceptable if boost dose is not possible due to clinical reasons or dosimetric constraints.
  2. Phase 2: (GTV only) Boost is not mandatory and up to the discretion of radiation oncologist. Total radiation prescription dose 5.4 Gy given in 3 fractions of 1.8 Gy per fraction, 5 fractions / week, one treatment .
  Arms: Neoadjuvant Chemoradiation

SUMMARY:
The best treatment for resectable esophageal or gastroesophageal adenocarcinoma is unknown. Although an operation to remove the esophagus is the most common treatment, previous studies have shown that patients live longer when either perioperative (before and after surgery) chemotherapy or preoperative (before surgery) chemotherapy plus radiation is given, compared to surgery alone. However it is unknown which of these treatments (perioperative chemotherapy or preoperative chemoradiation) is more effective in improving survival. A study where patients with resectable esophageal / GE junction cancer are chosen at random to receive one of the two preoperative treatments would help determine if one form of treatment improves survival compared to the other.

Patients with localized esophageal / GE junction cancer (adenocarcinoma) will be randomized to receive either preoperative and postoperative chemotherapy or preoperative chemoradiation followed by surgery.

The main objective of this pilot trial is to determine the possibility of conducting a larger study with many centers participating. If this study proves to be feasible with enough patients enrolled and able to tolerate treatments without major side effects then we can hopefully proceed to perform a larger multi-center trial to look for survival outcome differences between patients who receive preoperative chemotherapy and those who receive preoperative chemoradiation. The results of this trial would ultimately help us choose the most effective treatment of resectable esophageal cancer and hopefully improve survival.

DETAILED DESCRIPTION:
OBJECTIVE To determine the feasibility of a randomized trial of neoadjuvant chemotherapy vs. neoadjuvant chemoradiation for patients with resectable adenocarcinoma of the esophagus or gastroesophageal junction.

RESEARCH PLAN Phase III randomized 2-arm parallel group pilot study

1:1 randomization to A) or B)

TREATMENT REGIMEN A) PERIOPERATIVE CHEMOTHERAPY (OPTION of CHEMO REGIMEN 1 or 2) 1) FLOT - Four x 14 day cycles FLOT preoperatively and 4 cycles postoperatively: 5-Fluorouracil 2600 mg/m², day 1 IV every 14 days Leucovorin 200 mg/m², day 1, IV., every 14 days Oxaliplatin 85 mg/m², day 1, IV, every 14 days Docetaxel 50mg/m2, day 1, IV, every 14 days

OR

2) ECF / ECX - Three x 21-day cycles ECF preoperatively and 3 cycles postoperatively (within 4-10 weeks after surgery): Epirubicin (50 mg/m²,) day 1 IV Cisplatin: 60 mg/m², day 1 IV 5-Fluorouracil: 200 mg/m², daily for 21 days by continuous IV infusion 5-FU may be substituted with Capecitabine (Xeloda) 625mg/m2, BID (ECX)

OR

B) NEOADJUVANT CHEMORADIATION

1) -carboplatin and paclitaxel given on days 1, 8, 15, 22 and 29

* paclitaxel: 50 mg / m2 IV
* carboplatin: dosed to an area under the curve of 2, by Calvert formula Radiation Therapy 45-50.4 Gy in 25-28 fractions of 1.8 Gy/fraction, 5 fractions/wk 45-50.4 Gy in 25-28 fractions of 1.8 Gy/fraction, 5 fractions/wk Upon completion of neoadjuvant therapy, all patients will be considered for surgery.

Patients will be deemed acceptable for surgery provided:

* repeat imaging performed after neoadjuvant therapy does not demonstrate distant metastases or local invasion of the primary tumor into vital structures (heart, great vessels, trachea)
* maintenance of adequate performance status and ability to tolerate esophagectomy

Surgery will be performed preferably within 8 weeks of completion of neoadjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* adenocarcinoma of esophagus or gastroesophageal junction; -cT1N1-3 or T2-4Nx; M0 by American Joint Committee on Cancer (AJCC) 7th Edition staging classification
* proximal portion of the tumor at least 20 cm from the incisors on endoscopy, and extend no greater than 2 cm into the gastric cardia
* tumor length < 8cm; diameter < 5 cm
* age > 18 years
* absolute neutrophil count (ANC) ≥ 1.5 x 109 / L
* platelet count > 100 x 109 / L
* creatinine clearance > 50 ml / min
* bilirubin < 1.5x upper limit normal
* FEV1 > 1.0 L
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Exclusion Criteria

* positive serum / urine pregnancy test for females of childbearing age
* previous primary / recurrent malignancy in last 5 years (history of previous / current non-melanoma skin cancer or cervical in-situ carcinoma in last 5 years acceptable for inclusion in trial)
* previous chemotherapy for esophageal cancer
* previous radiation therapy that would overlap required radiation fields
* major systemic illness(es) that would limit life expectancy <2 years
* psychiatric / cognitive illness that would limit ability to give informed consent
* (Patients will be reviewed by both a medical and radiation oncologist and deemed fit to undergo either neoadjuvant chemotherapy or chemoradiation, respectively)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-08 (Actual); Study Completion 2023-08 (Actual)

PRIMARY OUTCOMES:
compliance with assigned neoadjuvant treatment | 5 weeks for chemoradiation arm, 6-8 weeks for chemotherapy arm
  - >60% patients allocated for randomization will start and complete treatment without major protocol violation
treatment response | 5 weeks for chemoradiation arm, 6-8 weeks for chemotherapy arm
  >30% of patients in both treatment arms demonstrate partial or complete response as defined by Mandard TRG 1-3 on pathologic staging

SECONDARY OUTCOMES:
survival | 3 years
  3 year overall- and disease-free survival
EORTC QOL | baseline, 3, 6, 9, 12 months post treatment
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C-30 Version 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Buduhan, MD MSc FRCSC, Principal Investigator — University of Manitoba / CancerCare Manitoba
Locations (3):
- Canada (3):
  - Health Sciences Centre / CancerCare Manitoba, Winnipeg, Manitoba
  - London Health Sciences Centre, London, Ontario
  - Toronto General Hospital / Princess Margaret Hospital, Toronto, Ontario